CLINICAL TRIAL: NCT04695171
Title: Cohort Registry on LINX Reflux Management System or Fundoplication Clinical Study in Patients With Hiatal Hernia >3 cm
Brief Title: LINX Reflux Management System or Fundoplication Clinical Study in Patients With Hiatal Hernia >3 cm
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early. The sponsor will focus on prospective randomized controlled studies at this time. Funding removed.
Sponsor: Foregut Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TRX-2019-02
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hiatal Hernia Large; Gastro Esophageal Reflux; Hiatal Hernia; Hiatal Hernia, Paraesophageal; Reflux, Gastroesophageal; Reflux Acid
Keywords: GERD; LINX; Fundoplication; MSA; Magnetic Sphincter Augmentation; MSAD; Magnetic Sphincter Augmentation Device
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal | interventions — Fundoplication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Prior Primary Large Hiatal Hernia with LINX Placement MSA: Patients who were previously implanted with the LINX device during repair of a hiatal hernia >3 cm >2 years prior will be asked to complete a quality of life questionnaire at about 3 years and 5 years post procedure. Each participant will complete a barium swallow at 3 and 5 years to determine recurrence of hiatal hernia.
  Interventions: Device: LINX Reflux Management System
- Prior Primary Large Hiatal Hernia with Fundoplication: Patients who previously underwent lower esophageal sphincter reconstruction by fundoplication during repair of a hiatal hernia >3 cm >2 years prior will be asked to complete a quality of life questionnaire at about 3 years and 5 years post procedure. Each participant will complete a barium swallow at about 3 and 5 years to determine recurrence of hiatal hernia.
  Interventions: Procedure: Fundoplication

INTERVENTIONS:
Device: LINX Reflux Management System — The LINX Reflux Management System consists of a series of titanium beads each with a magnetic core connected with independent titanium wires to form an annular shape when implanted. The attractive force of the magnetic beads is designed to provide additional strength to keep a weak lower esophageal sphincter (LES) closed. During swallowing, the magnetic beads slide away from each other on the independent titanium wire "links" to allow esophageal distention as the bolus passes by.
  Other Names: Magnetic Augmentation System; Magnetic Sphincter Augmentation Device, MSAD; Magnetic Sphincter Augmentation, MSA
  Groups: Prior Primary Large Hiatal Hernia with LINX Placement MSA
Procedure: Fundoplication — A surgical procedure where the fundus of the stomach is wrapped around and sutured to the distal esophagus to restore the function of the lower esophageal sphincter in limiting stomach contents from refluxing into the esophagus.
  Other Names: Nissen fundoplication; Partial fundoplication; Toupet fundoplication; Watson fundoplication; Dor fundoplication
  Groups: Prior Primary Large Hiatal Hernia with Fundoplication

SUMMARY:
The cohort registry is both retrospective and prospective, multicenter surveillance of subjects who underwent a prior hiatal hernia repair and Magnetic Sphincter Augmentation or fundoplication construction more than 2 years prior to initial study visit.

DETAILED DESCRIPTION:
The cohort registry is both retrospective and prospective, multicenter surveillance of subjects who underwent a prior hiatal hernia repair and anti-reflux surgery with either Magnetic Sphincter Augmentation (MSA) using LINX placement or fundoplication construction more than 2 years prior to initial study visit. Subjects will be enrolled by invitation only by participating investigators. Enrollment will consist of 300 LINX MSA patients and 150 fundoplication patients with a total of 450 from 4 sites within the United States. Data will be collected for up to 6 years.The primary objective of this study is to determine the long-term incidence of hiatal hernia recurrence in patients who undergo hiatal hernia repair of a large (>3 cm) hernia with LINX® device placement, and to compare this with hiatal hernia recurrence rates in patients who underwent hiatal hernia repair with fundoplication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 21 years of age and at least the minimum Age of Majority according to applicable state law.
2. Underwent primary index procedure of laparoscopic repair of a hiatal hernia larger than 3 cm with placement of a LINX® device or construction of a fundoplication for reflux control more than 2 years prior to his/her enrollment or has completed 1 or 2 of the barium swallows and GERD-HRQLs within study time points with or without hiatal hernia recurrence.
3. Subject is willing and able to cooperate with follow-up examinations.
4. Subject has been informed of the study procedures and treatment and has signed an informed consent.

Exclusion Criteria:

1. The surgical procedure was completed as an emergency procedure
2. Currently being treated with another investigational drug or investigational device
3. Suspected or confirmed esophageal or gastric cancer
4. Subject has Barrett's esophagus >3cm
5. Cannot understand trial requirements or is unable to comply with follow-up schedule
6. Pregnant or plans to become pregnant during the course of the study
7. Medical illness (i.e. congestive heart failure) that may cause the subject to be non-compliant with or able to meet the protocol requirements or is associated with limited life expectancy (i.e. less than 3 years)
8. Diagnosed psychiatric disorder (e.g. bipolar, schizophrenia, etc.), subjects that exhibit depression that are on appropriate medication(s) are allowable.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical evaluation will be conducted at four U.S. investigational centers with up to one hundred and fifty(150) subjects per center (goal of 450 total). Corhort 1 will consist of 300 subjects who were implanted with the LINX® Reflux Management System in the manner described above more than 2 years prior to enrollment to this study. Cohort 2 will consist of 150 subjects who underwent a fundoplication more that 2 years prior to enrollment into this study with similar hiatal hernia size and similar effective esophageal motility.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Hiatal Hernia Recurrence | Up to 5 years post index procedure
  The primary objective of this study is to determine the long-term incidence of hiatal hernia recurrence in patients who undergo primary hiatal hernia repair of a large (>3 cm) hernia with LINX® device placement, and to compare this with hiatal hernia recurrence rates in patients who undergo hiatal hernia repair with fundoplication.

SECONDARY OUTCOMES:
Incidence of Repeat Surgical Intervention | 5 years
  A secondary objectives are to determine the incidence of repeat surgical intervention with recurrent hernias in patients who received a LINX verses fundoplication.
Understanding Patient Reported Symptom Control | 5 years
  A secondary objective is to understand patient-reported symptom control including PPI use, occurrence rate of gas and bloating, and ability to belch and vomit as measured by comparison of pre- and post-operative satisfaction and ROARS Questionnaire (GERD-Health related quality of life [HRQL]) surveys during multiple follow-up time points.

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Bell, M.D., Principal Investigator — Principal Investigator
Locations (6):
- United States (6):
  - Keck Medical Center of USC, Los Angeles, California
  - Institute of Esophageal and Reflux Surgery, Lone Tree, Colorado
  - South Florida Reflux Center, Coral Springs, Florida
  - East Carolina University, Greenville, North Carolina
  - Esophageal Institute, Pittsburgh, Pennsylvania
  - University of Texas, Austin, Texas